CLINICAL TRIAL: NCT00927329
Title: Evaluation of the Safety and Effect of an Allergen Challenge Procedure on Nasal Airway Inflammation in Allergic Individuals Using a Dermatophagoides Farinae Extract Nasal Allergen Challenge Protocol
Brief Title: Evaluation of a Nasal Allergen Challenge Procedure Using Dust Mite Extract
Acronym: Dusty
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Original PI left institution.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 09-0196; 59719
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Dermatophagoides Farinae Allergy; Asthma; Healthy
Keywords: Dermatophagoides; farinae; allergen; dust; allergic; mite; allergy
MeSH Terms: conditions — Dust Mite Allergy; Asthma; Hypersensitivity | interventions — Sensitivity and Specificity; Anti-Allergic Agents; Allergens; Dust

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dust mite (Experimental)
  Interventions: Biological: dust mite inhalation

INTERVENTIONS:
Biological: dust mite inhalation — Nasal allergen challenge will be provided in a graded dose fashion of 0 AU, 100 AU, 500 AU, and 1000 AU separated by 20 minutes.
  Other Names: allergy; allergic; Dermatophagoides; farinae; allergen; dust allergy; dust; mite; mite allergy

SUMMARY:
The purpose of this study is to serve as a pilot safety study for nasal allergen challenges.

DETAILED DESCRIPTION:
The purpose of this study is to serve as a pilot safety study for the implementation of a new technique for nasal allergen challenges. The new technique consists of having patients maximally inhale to total lung capacity. A nasal metered dose pump will be used to deliver the Dermatophagoides farinae allergen to the nasal mucosa. The patient will not sniff after allergen delivery as in the previous study but instead exhale through the mouth. The investigators propose that this technique will inhibit large amounts of allergen reaching airway mucosa beyond the nasal site of introduction thus limiting serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Specific allergy to house dust mite Dermatophagoides farinae confirmed by positive immediate skin test response.
2. Subjects may be enrolled with mild asthma if they have an FEV1 of at least 80% of predicted and FEV1/FVC ratio of at least .70 (without the use of bronchodilating medications for 12 hours). This is consistent with lung function of persons with mild episodic or mild persistent asthma. For the purpose of this protocol, an asthmatic individual will be defined as having: a) a positive methacholine challenge with a provocative concentration of methacholine producing a 20% fall in FEV1 (PC20 methacholine) with less than or equal to 10 mg/ml by the method used; OR b) physician diagnosed asthma with symptoms and chronic daily therapy consistent with mild asthma.
3. Ability to withhold antihistamine medications for one week prior to screening visit and one week prior to nasal allergen challenge visit.
4. Subjects must be able and willing to give informed consent.

Exclusion Criteria:

1. Any chronic medical condition considered by the PI as a contraindication to the allergen challenge study including significant cardiovascular disease, diabetes requiring medication, chronic renal disease, or chronic thyroid disease.
2. Physician directed emergency treatment for an asthma exacerbation within the preceding 12 months.
3. Use of systemic steroid therapy within the preceding 12 months for treatment of an asthma exacerbation.
4. Use of inhaled or nasal steroids, cromolyn, or leukotriene inhibitors (Montelukast or Zafirlukast) within the past month (except for use of cromolyn exclusively prior to exercise).
5. Use of allergen immunotherapy.
6. Use of daily theophylline within the past month.
7. Use of nasal medications that might alter the response to nasal allergen challenge including anti-inflammatory and anti-histamine agents within one week of challenge.
8. Pregnancy or nursing a baby.
9. Cigarette smoking within the past 12 months.
10. Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
11. Exacerbation of asthma more than 2x/week which would be characteristic of a person with moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
12. Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma. (Not to include prophylactic use of albuterol prior to exercise).
13. Vitamin or herbal supplementation considered by the PI as having anti-inflammatory and/or anti-oxidant properties must be stopped 7 days prior to entrance into the study.
14. A history of nasal or sinus surgery within the last 5 years.
15. Viral URI within four weeks of challenge.
16. Acute infection requiring the use of antibiotics within the last four weeks. Must be off antibiotics for at least two weeks prior to study.
17. Participation in an allergen challenge study within two weeks of this challenge or use of an investigational agent within the last 30 days.
18. Use of tricyclic antidepressants, beta-blockers, monoamine oxidase inhibitors or other drugs that may interfere with the treatment of anaphylaxis.
19. Subjects with history of immunologic disease or on immune suppression for cancer or other disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01 (Estimated); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Successful nasal allergen challenge without serious adverse event. | Immediate

SECONDARY OUTCOMES:
analyze and compare cells of the airway and serum for a variety of inflammatory markers relevant to innate immunity. | 4 hr post exposure

CONTACTS AND LOCATIONS:
Overall Officials: David Peden, MD, Principal Investigator — University of North Carolina, Chapel Hill; Michelle Hernandez, MD, Study Director — University of North Carolina, Chapel Hill